CLINICAL TRIAL: NCT01950156
Title: Phase I/II Study Using Epitope Peptide Restricted to HLA-A*24 (URLC10,CDCA1,KIF20A) in Patients With Disease Controlled Advanced Non-small Cell Lung Cancer
Brief Title: Safety and Efficacy Study of Epitope Peptide To Treat HLA-A*24 Disease Controlled Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shiga University (Other)
Collaborators: Tokyo University (Other)
Responsible Party: Principal Investigator, Yataro Daigo, Professor, Shiga University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUMS-23-57; 23-57 (Other: Shiga University)
Record Dates: First submitted 2013-09-17; First posted 2013-09-25 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — NUF2 protein, human; Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (Experimental): HLA-A*2402restricted URLC10, CDCA1, and KIF20A peptides with adjuvant
  Interventions: Biological: HLA-A*2402restricted URLC10, CDCA1, and KIF20A peptides with adjuvant

INTERVENTIONS:
Biological: HLA-A*2402restricted URLC10, CDCA1, and KIF20A peptides with adjuvant — Open Label, Non-Randomized, Safety/Efficacy study: patients will be vaccinated subcutaneously once a week with HLA-A*2402restricted URLC10, CDCA1, and KIF20A peptides with adjuvant.

SUMMARY:
The investigators previously identified three novel HLA-A*2402-restricted epitope peptides, which were derived from three cancer-testis antigens, URLC10, CDCA1, and KIF20A, as targets for vaccination against lung cancer. In this clinical study, the investigators examine using a combination of these three peptides the safety, immunogenicity, and antitumor effect of vaccine treatment to prevent relapse of the disease for HLA-A*2402-positive advanced non-small cell lung cancer patients whose disease are controlled after any standard therapies.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, immune response and clinical efficacies of HLA-A*2402 restricted epitope peptides URLC10, CDCA1, and KIF20A emulsified with Montanide ISA 51 for disease controlled advanced non-small cell lung cancers.

The investigators previously identified three novel HLA-A*2402-restricted epitope peptides, which were derived from three cancer-testis antigens, URLC10, CDCA1, and KIF20A, as targets for cancer vaccination against lung cancer. In this phase I/II trial, the investigators examine using a combination of these three peptides the safety, immunogenicity, and antitumor effect of vaccine treatment for HLA-A*2402-positive advanced non-small cell lung cancer patients whose disease are controlled after any standard therapies, but who do not have any options for additional standard ones to prevent .future relapse of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. NSCLC whose disease are controlled after any standard therapies, but who do not have any additional standard ones to prevent .future relapse of the disease.
2. ECOG performance status 0-2
3. Age between 20 to 85
4. Clinical efficacy can be evaluated by some methods
5. No prior chemotherapy, radiation therapy, hyperthermia or immunotherapy within appropriate periods
6. Life expectancy > 3 months
7. Laboratory values as follows 1500/mm3 < WBC < 15000/mm3 Platelet count > 75000/mm3 Asparate transaminase < 3 X cutoff value Alanine transaminase < 3 X cutoff value Total bilirubin < 3 X cutoff value Serum creatinine < 2X cutoff value
8. HLA-A*2402
9. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Active and uncontrolled cardiac disease (i.e. coronary syndromes, arrhythmia)
2. Myocardial infarction within six months before entry
3. Breastfeeding and Pregnancy (woman of child bearing potential)
4. Active and uncontrolled infectious disease
5. Concurrent treatment with steroids or immunosuppressing agent
6. Other malignancy requiring treatment
7. Non-cured traumatic wound
8. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2011-09; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety: the number of adverse events of vaccination therapy. | 2 months
Evaluation of clinical efficacy: Progression free survival. | 2 months
Evaluation of clinical efficacy: Tumor markers. | 2 months
Evaluation of clinical efficacy: Overall survival. | 2 months
Evaluation of clinical efficacy: Objective response rate. | 2 months

SECONDARY OUTCOMES:
Various immunological responses comprising peptides specific CTL, antigen cascade, regulatory T cells, cancer antigens and HLA levels | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shiga University of Medical Science Hospital, Ōtsu, Shiga, Japan

REFERENCES:
- [Background] Kono K, Mizukami Y, Daigo Y, Takano A, Masuda K, Yoshida K, Tsunoda T, Kawaguchi Y, Nakamura Y, Fujii H. Vaccination with multiple peptides derived from novel cancer-testis antigens can induce specific T-cell responses and clinical responses in advanced esophageal cancer. Cancer Sci. 2009 Aug;100(8):1502-9. doi: 10.1111/j.1349-7006.2009.01200.x. Epub 2009 May 14. PMID 19459850
- [Background] Harao M, Hirata S, Irie A, Senju S, Nakatsura T, Komori H, Ikuta Y, Yokomine K, Imai K, Inoue M, Harada K, Mori T, Tsunoda T, Nakatsuru S, Daigo Y, Nomori H, Nakamura Y, Baba H, Nishimura Y. HLA-A2-restricted CTL epitopes of a novel lung cancer-associated cancer testis antigen, cell division cycle associated 1, can induce tumor-reactive CTL. Int J Cancer. 2008 Dec 1;123(11):2616-25. doi: 10.1002/ijc.23823. PMID 18770861
- [Background] Mizukami Y, Kono K, Daigo Y, Takano A, Tsunoda T, Kawaguchi Y, Nakamura Y, Fujii H. Detection of novel cancer-testis antigen-specific T-cell responses in TIL, regional lymph nodes, and PBL in patients with esophageal squamous cell carcinoma. Cancer Sci. 2008 Jul;99(7):1448-54. doi: 10.1111/j.1349-7006.2008.00844.x. Epub 2008 Apr 30. PMID 18452554
- [Background] Daigo Y, Nakamura Y. From cancer genomics to thoracic oncology: discovery of new biomarkers and therapeutic targets for lung and esophageal carcinoma. Gen Thorac Cardiovasc Surg. 2008 Feb;56(2):43-53. doi: 10.1007/s11748-007-0211-x. Epub 2008 Feb 24. PMID 18297458
- [Background] Ishikawa N, Takano A, Yasui W, Inai K, Nishimura H, Ito H, Miyagi Y, Nakayama H, Fujita M, Hosokawa M, Tsuchiya E, Kohno N, Nakamura Y, Daigo Y. Cancer-testis antigen lymphocyte antigen 6 complex locus K is a serologic biomarker and a therapeutic target for lung and esophageal carcinomas. Cancer Res. 2007 Dec 15;67(24):11601-11. doi: 10.1158/0008-5472.CAN-07-3243. PMID 18089789
- [Background] Suda T, Tsunoda T, Daigo Y, Nakamura Y, Tahara H. Identification of human leukocyte antigen-A24-restricted epitope peptides derived from gene products upregulated in lung and esophageal cancers as novel targets for immunotherapy. Cancer Sci. 2007 Nov;98(11):1803-8. doi: 10.1111/j.1349-7006.2007.00603.x. PMID 17784873
- [Background] Hayama S, Daigo Y, Kato T, Ishikawa N, Yamabuki T, Miyamoto M, Ito T, Tsuchiya E, Kondo S, Nakamura Y. Activation of CDCA1-KNTC2, members of centromere protein complex, involved in pulmonary carcinogenesis. Cancer Res. 2006 Nov 1;66(21):10339-48. doi: 10.1158/0008-5472.CAN-06-2137. PMID 17079454